CLINICAL TRIAL: NCT04686188
Title: Exploring the Mechanisms and Dynamics of Clonal Evolution Leading to Recurrence in Prostate Cancer Through Evaluation of Intratumour Heterogeneity at Diagnosis and Circulating Tumour DNA at Recurrence
Brief Title: Exploring the Mechanisms and Dynamics of Clonal Evolution Leading to Recurrence in Prostate Cancer
Acronym: EXCERPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5314; 275583 (Other: NHS Health Research Authority)
Record Dates: First submitted 2020-12-10; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer Recurrent
Keywords: Prostate cancer; Liquid biopsy; Circulating tumor DNA; Intratumor Heterogeneity; Prostate radiotherapy; Recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample(s) to be collected from patients and then stored under unique trial identifier in the Principal Investigator's laboratory at the Institute of Cancer Research. Samples to be collected for DNA extraction, library prep, sequencing, and bioinformatic analysis. Remaining biological material to be sent to ICR Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer is the most common cancer in males in the UK, and current estimates are that 1 in 8 will be diagnosed with prostate cancer in their lifetime. Although surgery or radiotherapy with hormone therapy offers a good chance of cure in localised disease, recurrence can occur, which may cause significant distress, and may shorten the patient's life. In patients with locally advanced disease (disease that has broken through the surrounding capsule of the prostate gland), around 30-40% of patients experience a recurrence.

Cancer develops as a result of normal cells acquiring genetic mutations, and localised prostate cancer at diagnosis is commonly made up of different subclones - distinct regions within the patient's cancer with different sets of genetic mutations, each of which may behave differently and be more or less sensitive to treatments.

The IMRT clinical trial (CCR 1766) recruited 486 patients who received hormone therapy and radiotherapy to the prostate and lymph nodes in patients with locally advanced prostate cancer. The FORECAST study (FORecasting the Evolution of CAncer of the proState within a Trial) is undertaking genetic sequencing of several regions of these patients' prostate cancers in order to determine which subclones are present at diagnosis, and how they evolved. FORECAST also has permission to obtain and perform sequencing on primary samples from two other large trials in localized prostate cancer.

This study seeks to collect blood samples from patients who have experienced a recurrence in whom the primary biopsies have been sequenced as part of FORECAST. Additionally, blood will be collected from any patient in follow up at The Royal Marsden who received radiotherapy and hormone therapy for a localised prostate cancer and has experienced a recurrence but not yet started treatment. In these patients, the FORECAST protocol will be used to undertake genetic sequencing of their original prostate cancer biopsies. Genetic mutations from the cancer can be detected in the blood in patients who relapse, so-called 'liquid biopsies'. By comparing the genetic information between the primary and relapsed cancer, we can detect which subclones present at diagnosis are ultimately responsible for the cancer relapsing, and help us to understand the evolution of prostate cancers over time. This will assist us in predicting at the point of diagnosis which patients are more likely to relapse, so that we may consider escalating primary treatments or treating patients with high-risk subclonal mutations with targeted therapies upfront. As a result, we aim to reduce the number of patients treated for localised prostate cancer experiencing a recurrence. Additionally, although liquid biopsies are well-characterized in metastatic prostate cancer, little is known about their value in patients who have a biochemical-only relapse (patients who have a rising PSA with no evidence of cancer on scans) and this will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged ≥18 years
2. Prostate tumour biopsy specimens available at The Royal Marsden Hospital, Kingston Hospital, Epsom and St Helier Hospitals, St George's Hospital or Croydon University Hospital and >2 primary tumour regions sampled
3. Received primary radical radiotherapy and androgen deprivation therapy and remains under follow up at The Royal Marsden Hospital
4. Willing and able to comply with blood sample collection
5. Capable of understanding and complying with the protocol requirements and has given written, dated and signed informed consent AND
6. Confirmed biochemical or radiological evidence of recurrent prostate cancer, and not yet received treatment for recurrent disease OR
7. FORECAST patients with confirmed biochemical or radiological evidence of recurrent prostate cancer who have received or are currently receiving treatment but are progressing (rising PSA and/or evidence of progressive disease on imaging), or have a PSA >2ng/ml

Exclusion Criteria:

1. Patients who have had another malignancy (excluding non-melanoma skin cancer, in-situ or superficial bladder cancer) treated within the previous 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient prostate cancer follow up clinics at the Royal Marsden Hospital in Sutton, England.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the evolution of prostate cancers from localised disease to recurrence | Until completion of study - predicted date 1 Sept 2022
  This is a basic science/ translational study and therefore no strict pre-determined primary outcome can be defined as it is hypothesis-generating. This study aims to identify prognostic evolutionary or genetic biomarkers in localised prostate cancers and such biomarkers can then be evaluated further in clinical studies.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sottoriva, BSc MSc PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Fully anonymised DNA sequencing data will be stored in an online repository such as the European Genome- Phenome Archive at the European Bioinformatics Institute, or the forthcoming ICR (Institute of Cancer Research) repository. The data will be encrypted and accessible only to us unless a potential collaborator enters into an agreement with our group at the ICR and we agree to share the data as part of an ethically-approved study. No patient-identifiable information will be shared.